CLINICAL TRIAL: NCT01253824
Title: Pharmacodynamics of NPC-01( 1mg Norethisterone and 0.02mg Ethinyl Estradiol) and IKH-01( 1mg Norethisterone and 0.035mg Ethinyl Estradiol); Effect of NPC-01 and IKH-01 on Serum Concentrations of Estradiol, Progesterone, FSH and LH.
Brief Title: Pharmacodynamics of NPC-01/IKH-01; Effect of NPC-01/IKH-01 on Sexual Hormone Concentrations in Healthy Female Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPC-01-4
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: NPC-01; IKH-01; Pharmacodynamics; Norethisterone; Ethinyl Estradiol; Estradiol; Progesterone; FSH; LH
MeSH Terms: interventions — Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPC-01 (Experimental): 1mg norethisterone and 0.02mg ethinyl estradiol
  Interventions: Drug: NPC-01
- IKH-01 (Active Comparator): 1mg norethisterone and 0.35mg ethinyl estradiol
  Interventions: Drug: IKH-01

INTERVENTIONS:
Drug: NPC-01 — NPC-01 contains 1mg norethisterone and 0.02mg ethinyl estradiol
  Other Names: norethisterone and ethinyl estradiol
  Arms: NPC-01
Drug: IKH-01 — IKH-01 contains 1mg norethisterone and 0.35mg ethinyl estradiol
  Other Names: norethisterone and ethinyl estradiol
  Arms: IKH-01

SUMMARY:
The purpose of this study is to compare the serum levels of estradiol, progesterone, FSH and LH in NPC-01 or IKH-01 one treatment cycle with those in before and after administration cycle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female aged between 20 to 35 years
* BMI:18.0-26.0

Exclusion Criteria:

* Females who are pregnant
* Drug use affecting sex hormone secretion

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takefumi Matuo, MD, Principal Investigator — Hyogo Prefectural AWAJI Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty one subjects were screened for this study after acquiring an informed consent.
  18 subjects of those participated in pre-medication menstrual cycle phase to confirm baseline of estradiol, progesterone, FSH and LH.
  4 subjects withdrew IC during this phase, therefore, 14 subjects were registered and allocated study drugs.
Period: Overall Study
Arm/Group | NPC-01 | IKH-01
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects were included for safety and pharmacodynamics analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | NPC-01 | IKH-01 | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (2.3) | 26.1 (4.4) | 26.4 (3.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 7 | 7 | 14
Body weight [Mean (Standard Deviation); unit: kg] | 51.14 (4.23) | 51.86 (6.03) | 51.5 (5.01)

OUTCOME MEASURES:

1. Primary Outcome: Comparing Estradiol AUC of Menstrual Period During Study Drug Administration With Pre and Post Study Drug Administration (Baseline(BL)-Study Drug Administration(SDA), Follow up(FU)-Study Drug Administration(ADA))
Description: Estradiol was measured on day 3, 6, 9, 12, 15, 18, 21, 24 on 3 consecutive menstrual period (pre administration/Baseline(BL), study drug administration(SDA), post administration/follow up(FU)) and calculated AUC from these data
Time Frame: Day 3, 6, 9, 12, 15, 18, 21, 24 of menstrual cycles
Measure: Mean (Standard Deviation); unit: pg･day/mL,
Arm/Group | NPC-01 | IKH-01
Number analyzed (Participants) | 7 | 7
pg･day/mL,
  Difference of estradiol AUC (BL-SDA) | 1654.7 (1652.6) | 2478.0 (793.0)
  Difference of estradiol AUC(FU-SDA) | 1872.6 (1819.2) | 2434.9 (1151.5)

2. Secondary Outcome: Comparing FSH AUC of Menstrual Period During Study Drug Administration With Pre and Post Study Drug Administration (Baseline(BL)-Study Drug Administration(SDA), Follow up(FU)-Study Drug Administration(ADA))
Description: FSH was measured on day 3, 6, 9, 12, 15, 18, 21, 24 on 3 consecutive menstrual period (pre administration/Baseline(BL), study drug administration(SDA), post administration/follow up(FU)) and calculated AUC from these data
Time Frame: Day 3, 6, 9, 12, 15, 18, 21, 24 of menstrual cycles
Measure: Mean (Standard Deviation); unit: mIU･day/mL
Arm/Group | NPC-01 | IKH-01
Number analyzed (Participants) | 7 | 7
mIU･day/mL
  Differnce of FSH (BL-SDA) | -9.609 (20.879) | -4.380 (18.034)
  Difference of FSH(FP-SDA) | -4.404 (41.309) | 0.538 (30.497)

3. Primary Outcome: Comparing Progesterone AUC of Menstrual Period During Study Drug Administration With Pre and Post Study Drug Administration (Baseline(BL)-Study Drug Administration(SDA), Follow up(FU)-Study Drug Administration(ADA))
Description: Progesterone was measured on day 3, 6, 9, 12, 15, 18, 21, 24 on 3 consecutive menstrual period (pre administration/Baseline(BL), study drug administration(SDA), post administration/follow up(FU)) and calculated AUC from these data
Time Frame: Day 3, 6, 9, 12, 15, 18, 21, 24 of menstrual cycles
Measure: Mean (Standard Deviation); unit: ng･day/mL
Arm/Group | NPC-01 | IKH-01
Number analyzed (Participants) | 7 | 7
ng･day/mL
  Difference of progesterone(BL-SDA) | 54.171 (25.769) | 93.148 (45.867)
  Difference of progesterone(FU-SDA) | 89.711 (47.882) | 59.344 (49.160)

4. Secondary Outcome: Comparing LH AUC of Menstrual Period During Study Drug Administration With Pre and Post Study Drug Administration (Baseline(BL)-Study Drug Administration(SDA), Follow up(FU)-Study Drug Administration(ADA))
Description: LH was measured on day 3, 6, 9, 12, 15, 18, 21, 24 on 3 consecutive menstrual period (pre administration/Baseline(BL), study drug administration(SDA), post administration/follow up(FU)) and calculated AUC from these data
Time Frame: Day 3, 6, 9, 12, 15, 18, 21, 24 of menstrual cycles
Measure: Mean (Standard Deviation); unit: mIU･day/mL
Arm/Group | NPC-01 | IKH-01
Number analyzed (Participants) | 7 | 7
mIU･day/mL
  Difference of LH(BL-SDA) | 60.874 (41.200) | 57.124 (50.821)
  Difference of LH(FU-SDA) | 61.571 (89.546) | 59.837 (25.549)

ADVERSE EVENTS:
Arm/Group | NPC-01 | IKH-01
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPC-01 (N=7) | IKH-01 (N=7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 5 (6) | 3 (8)
Oligomenorrhoea (Reproductive system and breast disorders) | 2 (3) | 4 (4)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Plasminogen increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the sponsor and PI that no restricts the PI's right but need to discuss the timing of publish date of trial results after the trial is completed.